CLINICAL TRIAL: NCT06428409
Title: A Phase 1/2 Study to Evaluate the Safety and Efficacy of MK-2870 Monotherapy or in Combination With Other Anticancer Agents in Gastrointestinal Cancers
Brief Title: A Clinical Study of MK-2870 Alone or With Other Treatments to Treat Gastrointestinal Cancers (MK-9999-02A)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9999-02A; MK-9999-02A (Other: MSD); 2023-508703-21-00 (Registry Identifier: EU CT); U1111-1298-8273 (Registry Identifier: UTN); jRCT2031240178 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Pancreatic Ductal Adenocarcinoma; Biliary Tract Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Biliary Tract Neoplasms | interventions — Fluorouracil; Leucovorin; Levoleucovorin; Cisplatin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sacituzumab tirumotecan + Chemotherapy (Experimental): Participants will receive sacituzumab tirumotecan in one of two dose levels and chemotherapy every 2 weeks (Day 1 and Day 15 of every 4-week cycle). Participants will continue to receive the treatment until the cancer gets worse or they don't tolerate treatment.
  Interventions: Biological: Sacituzumab tirumotecan; Drug: Fluorouracil (5-FU); Drug: Leucovorin (LV) or levoleucovorin; Drug: Rescue medication; Drug: Supportive care measures
- Sacituzumab tirumotecan (Experimental): Participants will receive sacituzumab tirumotecan in one of two dose levels every 2 weeks (Day 1 and Day 15 of every 4-week cycle). Participants will continue to receive the treatment until the cancer gets worse or they don't tolerate treatment.
  Interventions: Biological: Sacituzumab tirumotecan; Drug: Rescue medication; Drug: Supportive care measures
- Sacituzumab tirumotecan + Cisplatin + Pembrolizumab (Experimental): Participants will receive sacituzumab tirumotecan in one of two dose levels on Day 1 and Day 8 of every 3-week cycle until the cancer gets worse or they don't tolerate treatment, cisplatin on Day 1 and Day 8 of each 3-week cycle for up to 8 cycles (up to approximately 6 months), and pembrolizumab on Day 1 of each 3-week cycle for up to approximately 2 years.
  Interventions: Biological: Sacituzumab tirumotecan; Drug: Rescue medication; Drug: Supportive care measures; Drug: Cisplatin; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Sacituzumab tirumotecan — Given by IV infusion.
  Other Names: MK-2870; SKB264
Drug: Fluorouracil (5-FU) — 5-FU is administered by IV infusion over 46 to 48 hours every 2 weeks.
  Arms: Sacituzumab tirumotecan + Chemotherapy
Drug: Leucovorin (LV) or levoleucovorin — LV or levoleucovorin is administered by IV infusion every 2 weeks.
  Arms: Sacituzumab tirumotecan + Chemotherapy
Drug: Rescue medication — Participants receive the following rescue medications, per approved product label, as premedication to study treatment to prevent hypersensitivity and/or infusion reactions: diphenhydramine (or equivalent histamine-1 [H1] receptor antagonist), H2 receptor antagonist, acetaminophen or equivalent, and dexamethasone or equivalent infusion. A steroid mouthwash (dexamethasone or equivalent) will be given as prophylaxis for stomatitis/oral mucositis.
Drug: Supportive care measures — Participants are allowed to take supportive care measures for the management of adverse events associated with study intervention at the discretion of the investigator. Supportive care measures may include but are not limited to antidiarrheal agents and antiemetic agents. Artificial tear drops or gel may be given as supportive care for Ocular Surface Toxicity.
Drug: Cisplatin — Given by IV infusion.
  Other Names: PLATINOL®
  Arms: Sacituzumab tirumotecan + Cisplatin + Pembrolizumab
Biological: Pembrolizumab — Given by IV infusion.
  Other Names: MK-3475; KEYTRUDA®
  Arms: Sacituzumab tirumotecan + Cisplatin + Pembrolizumab

SUMMARY:
Researchers want to learn if sacituzumab tirumotecan (MK-2870) alone or with other treatments can treat certain gastrointestinal (GI) cancers. The GI cancers being studied are either advanced (the cancer has spread to other parts of the body), or unresectable (the cancer cannot be removed with surgery). The goals of this study are to learn:

* About the safety of sacituzumab tirumotecan alone or with other treatments and if people tolerate it
* How many people have the cancer respond (get smaller or go away) to treatment

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has one of the following cancers:

  * Unresectable or metastatic colorectal cancer and has received prior therapy for the cancer
  * Advanced or metastatic pancreatic ductal adenocarcinoma (PDAC) and has received prior therapy for the cancer
  * Advanced and/or unresectable biliary tract cancer (BTC) and has received prior therapy for the cancer
  * Advanced and/or unresectable BTC and has not received prior therapy for the cancer
* For participants who have received prior therapy for cancer: Has recovered from any side effects due to previous cancer treatment

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* History of severe eye disease
* For participants who have received prior therapy for cancer: Received prior systemic anticancer therapy including investigational agents within 4 weeks before starting study intervention
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2029-10-16 (Estimated); Study Completion 2029-10-16 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience a Dose-limiting Toxicity (DLT) | Up to approximately 4 weeks
  A DLT is a medical problem related to the study medicine that prevents giving participants a higher dose or may prevent giving the participant the same dose. The number of participants who experience a DLT will be reported.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 63 months
  An AE is a health problem that happens or worsens during the study. The number of participants who have an AE during the study will be reported.
Number of Participants who Discontinue Study Treatment due to an AE | Up to approximately 63 months
  An AE is a health problem that happens or worsens during a study. The number of participants who stop study treatment will be reported.
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 63 months
  ORR is defined as the percentage of participants with confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.

SECONDARY OUTCOMES:
Duration of Response (DOR) per RECIST 1.1 as Assessed by BICR | Up to approximately 63 months
  For participants who demonstrate a confirmed Complete Response or Partial Response, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Progression-free Survival (PFS) per RECIST 1.1 as Assessed by BICR | Up to approximately 63 months
  PFS is defined as the time from start of study treatment to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. According to RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Overall Survival (OS) | Up to approximately 63 months
  OS is the length of time from when the participant starts treatment until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (55):
- United States (13):
  - UCLA ( Site 0317), Los Angeles, California
  - University of Colorado Anschutz Medical Campus ( Site 0299), Aurora, Colorado
  - University of Colorado Anschutz Medical Campus ( Site 0325), Aurora, Colorado
  - University of Colorado Anschutz Medical Campus ( Site 0326), Aurora, Colorado
  - Sibley Memorial Hospital ( Site 0310), Washington D.C., District of Columbia
  - University of Florida College of Medicine ( Site 0281), Gainesville, Florida
  - Mount Sinai Cancer Center ( Site 0287), Miami Beach, Florida
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital ( Site 0303), Marietta, Georgia
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island ( Site 0327), Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone ( Site 0324), New York, New York
  - University of Texas MD Anderson Cancer Center ( Site 0316), Houston, Texas
  - Oncology and Hematology Associates of Southwest Virginia (BRCC) ( Site 0295), Roanoke, Virginia
  - University Hospital and UW Health Clinics-Carbone Cancer Center ( Site 0293), Madison, Wisconsin
- Australia (5):
  - Westmead Hospital ( Site 0003), Westmead, New South Wales
  - Royal Brisbane and Women's Hospital-Medical Oncology Clinical Trials Unit, Cancer Care Services ( Site 0001), Brisbane, Queensland
  - Epworth Freemasons ( Site 0005), East Melbourne, Victoria
  - Frankston Hospital-Oncology and Haematology ( Site 0004), Frankston, Victoria
  - One Clinical Research ( Site 0002), Nedlands, Western Australia
- Canada (3):
  - The Ottawa Hospital Cancer Centre ( Site 0027), Ottawa, Ontario
  - Centre Hospitalier de l'Université de Montréal-Unit for Innovative Therapies ( Site 0022), Montreal, Quebec
  - McGill University Health Centre ( Site 0023), Montreal, Quebec
- Chile (4):
  - FALP-UIDO ( Site 0041), Providencia, Region M. de Santiago
  - Clínica UC San Carlos de Apoquindo ( Site 0043), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0047), Santiago, Region M. de Santiago
  - James Lind Centro de Investigacion del Cancer ( Site 0048), Temuco, Región de la Araucanía
- China (6):
  - Beijing Cancer hospital-Digestive Oncology ( Site 0061), Beijing, Beijing Municipality
  - The 900th Hospital of the Joint Logistics Support Force of the Chinese People's Liberation Army ( Site 0063), Fuzhou, Fujian
  - Wuhan Union Hospital Cancer Center. ( Site 0064), Wuhan, Hubei
  - Hunan Cancer Hospital-intervention department ( Site 0066), Changsha, Hunan
  - Renji Hospital Shanghai Jiao Tong University School of Medicine-Oncology Department ( Site 0067), Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University ( Site 0068), Chengdu, Sichuan
- Italy (3):
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 0101), Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda ( Site 0102), Milan, Lombardy
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -Medical Oncology ( Site 0103), Roma
- Japan (2):
  - National Cancer Center Hospital East ( Site 0121), Kashiwa, Chiba
  - Kanagawa Cancer Center ( Site 0122), Yokohama, Kanagawa
- South Korea (4):
  - Seoul National University Hospital ( Site 0161), Seoul
  - Severance Hospital, Yonsei University Health System ( Site 0164), Seoul
  - Asan Medical Center ( Site 0163), Seoul
  - Samsung Medical Center ( Site 0162), Seoul
- Spain (3):
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON-ONCOLOGY ( Site 0183), Madrid, Madrid, Comunidad de
  - Hospital Universitario Central de Asturias-Medical Oncology ( Site 0182), Oviedo, Principality of Asturias
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 0181), Barcelona
- Switzerland (2):
  - Hôpitaux Universitaires de Genève (HUG) ( Site 0202), Geneva, Canton of Geneva
  - Ospedale Regionale Bellinzona e Valli ( Site 0201), Bellinzona, Canton Ticino
- Taiwan (5):
  - China Medical University Hospital ( Site 0223), Taichung
  - National Cheng Kung University Hospital-Clinical Trial Center ( Site 0224), Tainan
  - National Taiwan University Hospital-Oncology ( Site 0225), Taipei
  - Taipei Veterans General Hospital ( Site 0221), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 0222), Taoyuan District
- Turkey (Türkiye) (2):
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 0241), Ankara
  - Ankara Bilkent Şehir Hastanesi-Medical Oncology ( Site 0242), Ankara
- United Kingdom (3):
  - Barts Health NHS Trust ( Site 0263), London, England
  - Royal Free Hospital ( Site 0262), London, England
  - University Hospital Coventry & Warwickshire ( Site 0266), Coventry

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26293&tenant=MT_MSD_9011